CLINICAL TRIAL: NCT01507285
Title: A Randomised, Double-blind, Placebo-controlled, Dose-escalation, Parallel-group, Single and Multiple Dosing Trial of NN90-1170 in Healthy Volunteers and Patients With Type 2 Diabetes to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics
Brief Title: Safety and Tolerability of Liraglutide in Healthy Volunteers and Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1189
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC 90-1170 (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Initial single dose followed by subsequent multiple s.c. (under the skin) doses on several dose levels (1.25, 5, 7.5, 10 and 12.5 mcg/kg). Each subject will be allocated to one dose level only
  Other Names: NNC 90-1170
  Arms: NNC 90-1170
Drug: placebo — Initial single dose followed by subsequent multiple s.c. (under the skin) doses
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess the safety and tolerability (maximum tolerated dose) after single and multiple doses of NNC 90-1170 (liraglutide) in healthy volunteers and in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HEALTHY VOLUNTEERS
* Healthy subjects aged 18-45 years inclusive
* Healthy subjects are defined as individuals free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, neurological and psychiatric disease as determined by history, physical examination and clinical laboratory test results
* Women who are not of childbearing potential
* Signed and dated written informed consent obtained
* Body mass index (BMI) within the range 19-30 kg/m^2, inclusive
* SUBJECTS WITH DIABETES
* Subjects aged 40-70 years inclusive
* Subjects diagnosed with type-2 diabetes and a duration of diabetes of more than 12 months
* Women who are not of childbearing potential
* Signed and dated written informed consent obtained
* Fasting C-peptide at least 0.3 nmol/l and blood glucose at least 7 mmol/l
* Subjects currently on diet and/or OHA (oral hypoglycemic agents) for at least six months
* Body mass index (BMI) below 35 kg/m^2
* HbA1c (glycosylated haemoglobin) below 11%
* Stable on current medication for at least 3 weeks prior to dosing in this study

Exclusion Criteria:

* HEALTHY VOLUNTEERS
* Clinically relevant abnormal history or physical findings (e.g. cancer) at the screening assessment, which could interfere with the objectives of the study or the safety of the subject's participation
* Clinically relevant abnormalities of laboratory values or ECG at the screening evaluation
* Presence of acute or chronic illness sufficient to invalidate the subject's participation in the study or to make it unnecessarily hazardous
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-150 mmHg systolic, 40-90 mmHg diastolic: heart rate 40-100 beats/min
* History of drug or alcohol abuse (alcohol abuse is defined as intake of more than 28 units weekly in men and more than 21 units weekly in women)
* Alcohol intake within 48 hours prior to visit
* Evidence of drug abuse on urine testing at study entry
* The subject smokes 10 cigarettes or more, or the equivalent, per day and is unable to refrain from smoking during 3 days prior to the first dosing day and during the confinement period
* Hepatitis B surface antigen (HBsAg), Hepatitis C antibodies or HIV (human immunodeficiency virus) antibodies
* History of significant drug allergy or drug hypersensitivity
* SUBJECTS WITH DIABETES
* Use of any drug (except for oral hypoglycaemic agents (OHAs)) which in the Investigator's opinion could interfere with the blood glucose level (e.g. insulin, systemic corticosteroids, thiazides)
* Recurrent severe hypoglycaemia as judged by the Investigator
* Clinically relevant abnormal history or physical findings (e.g. cancer) at the screening assessment, which could interfere with the objectives of the study or the safety of the subject's participation
* Clinically relevant abnormalities of laboratory values or ECG at the screening evaluation
* Presence of acute or chronic illness sufficient to invalidate the subject's participation in the study or to make it unnecessarily hazardous
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 110-160 mmHg systolic, 60-90 mmHg diastolic: heart rate 40-100 beats/min
* History of drug or alcohol abuse (alcohol abuse is defined as intake of more than 28 units weekly in men and more than 21 units weekly in women)
* Alcohol intake within 48 hours of visit
* Evidence of drug abuse on urine testing at study entry
* The subject smokes 10 cigarettes or more, or the equivalent, per day and is unable to refrain from smoking during 3 days prior to the first dosing day and during the confinement period
* Hepatitis B surface antigen (HBsAg), Hepatitis C antibodies
* History of significant drug allergy or drug hypersensitivity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1999-08; Primary Completion 1999-11 (Actual); Study Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Area under the Curve

SECONDARY OUTCOMES:
Cmax, maximum concentration
tmax, time to maximum concentration
t½, terminal half-life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manchester, United Kingdom

REFERENCES:
- [Result] Agerso H, Jensen LB, Elbrond B, Rolan P, Zdravkovic M. The pharmacokinetics, pharmacodynamics, safety and tolerability of NN2211, a new long-acting GLP-1 derivative, in healthy men. Diabetologia. 2002 Feb;45(2):195-202. doi: 10.1007/s00125-001-0719-z. PMID 11935150
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com